CLINICAL TRIAL: NCT02289248
Title: Cognitive Behavioral Therapy in Prolonging the Antidepressant Effects of Intravenous Ketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1501015171
Record Dates: First submitted 2014-11-04; First posted 2014-11-13 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Ketamine; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine/CBT Group (Experimental): Subjects will undergo 2 week course of 4 intravenous infusions of ketamine (given twice weekly for two weeks) in combination with twice weekly cognitive behavioral therapy for a total of 8 weeks.
  Interventions: Drug: Ketamine; Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Drug: Ketamine — Subjects will undergo a twice weekly two week course of IV infusions of ketamine
Behavioral: Cognitive Behavioral Therapy (CBT) — Subjects will undergo twice weekly CBT for a total of 8 weeks

SUMMARY:
Subjects with depressive episodes will be recruited to undergo a brief 2 week course of IV infusions of ketamine in combination with cognitive behavioral therapy for 8 weeks.

DETAILED DESCRIPTION:
Twelve subjects with current diagnosis of depressive episode will be recruited to undergo a brief course of 4 intravenous infusions of ketamine, given twice weekly for two weeks in combination with CBT, given twice weekly. The CBT course will be 16 total sessions (given over 8 weeks), will begin the day following the initial ketamine infusion, and will be performed by a therapist who has successfully completed extensive training at the Beck Institute for Cognitive Therapy and Research and has experience with similar studies. Homework assignments will include thought records and activity charts which are used in standard practice to facilitate CBT interventions.

ELIGIBILITY:
Inclusion Criteria:

* suffering from a depressive episode (DSM 5; either Major Depressive Disorder or Bipolar Disorder) and having failed one or more standard antidepressant treatments during the current episode;
* Age 18-65;
* Hamilton Depression Rating Scale (17-HAM-D) score of 21 or more prior to study entry.

Exclusion Criteria:

* Any Axis I or Axis II Disorder, which at screening is clinically predominant to their depressive episode or has been predominant to their depressive episode at any time within 6 months prior to screening;
* Active suicidal thoughts with a plan; current or recent (<6 months ago) substance use disorder;
* Non-affective psychosis (such as schizophrenia or schizoaffective disorder);
* Pregnancy or breastfeeding;
* Inability to speak English fluently;
* A clinically significant abnormality on the screening physical examination that might affect safety, study participation, or confound interpretation of study results;
* A history of CBT treatment in the past 12 months;
* Dementia;
* Delirium;
* Any other neurological or mental disease that might affect cognition or the ability to meaningfully participate in CBT.
* Untreated hypertension as defined by a systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg at screening on two of three measurements.
* Recent myocardial infarction (within one year)
* Syncopal event within the past year.
* Congestive heart failure (CHF) New York Heart Association Criteria >Stage 2
* Angina pectoris.
* Heart rate <50 or >105 beats per minute at screening

Females are eligible provided they meet criteria A or B below:

1. Non-childbearing potential: e.g., physiologically incapable of becoming pregnant, i.e., permanently sterilized (status post hysterectomy, bilateral tubal ligation), or is post-menopausal with her last menses at least one year prior to screening; or
2. Childbearing potential, and meets the following criteria:

i. Childbearing potential, including women using any form of hormonal birth control, on hormone replacement therapy started prior to 12 months of amenorrhea, using an intrauterine device (IUD), having a monogamous relationship with a partner who has had a vasectomy, or is sexually abstinent.

ii. Negative urinary pregnancy test at screening, confirmed by a negative urinary pregnancy test at enrollment prior to receiving study treatment.

iii. Willing and able to continuously use one of the following methods of birth control during the course of the study, defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly: implants, injectable or patch hormonal contraception, oral contraceptives, IUD, double-barrier contraception, sexual abstinence. The form of birth control will be documented at screening and baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-02; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Extinction Learning Task performance | 24 hours Post ketamine infusion
  Hopkins Verbal Learning Test and extinction learning tasks will be administered both one week before and 24-hours after the first ketamine infusion and the change in scores compared.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks
  Change in MADRS from baseline through week eight using a random effects model

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Wilkinson, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale Psychiatric Hospital, New Haven, Connecticut